CLINICAL TRIAL: NCT04956055
Title: The Effect of Hand Reflexology on Anxiety and Vital Signs in Patients With Coronary Angiography
Brief Title: The Effect of Hand Reflexology on Anxiety and Vital Signs With Angiography
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 16.03.2020-35
Record Dates: First submitted 2021-03-28; First posted 2021-07-09 (Actual); Last update posted 2021-07-09 (Actual); Status verified 2021-01

CONDITIONS: Coronary Artery Disease; Coronary Disease
Keywords: anxiety; life findings; coronary angiography; distress; reflexology; angiography
MeSH Terms: conditions — Coronary Artery Disease; Coronary Disease; Anxiety Disorders | interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Intervention Model Description: Single blind randomized controlled trial
Who Masked: Participant
Masking Description: Patients
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experiment group (Experimental): Experimental group to be applied hand reflexology
  Interventions: Other: Reflexology
- Control group (No Intervention): experimental group for which hand reflexology will not be applied

INTERVENTIONS:
Other: Reflexology — The patient will be kept in a lying position. First, the patient will be given four minutes of hand reflexology on each hand with warming and stimulation techniques.Reflexology will be applied to the left hand with the thumb of the right hand, the thumb of the left hand and the special points in the right hand. It will be applied to the fingers, palm, back of the hand, and finally the wrists, respectively, starting with the fingertips and using special reflexology techniques (a total of six minutes for each hand separately). By sending a moderate stimulus, a total of 20 minutes of reflexology session will continue.Since the patient reveals and uses his own internal energy at the end of the session, nobody should talk to the patient until five minutes after the procedure. Survey questions and vital signs would be examined five minutes after the session and the research with the participant would end.
  Arms: Experiment group

SUMMARY:
This study was planned to determine the effect of hand reflexology on anxiety and vital signs in patients undergoing coronary angiography. In the G-power analysis conducted to determine the sample of the study, experiment and control were calculated as 60 in total, with the sample number of both groups being 30. Since the study is a single-blind randomized clinical trial, in order to determine the randomization , a box with the names of the patients determined according to the participation criteria will be determined by the selection of the healthcare personnel responsible for the service, and the experimental and control groups. "Demographic Data Form" , "Distress Thermometer". "State Anxiety Inventory" , "Vital Signs Form" and Visual Analog Scale will be used to collect research data.

DETAILED DESCRIPTION:
Reflexology is a technique of pressure or pressure that is applied manually to the special points of the hand, foot and sometimes ear areas. Reflexology is applied to the soles of the hands and feet, its circumference, surface, inner and outer edges and the ear area The most important differences that distinguish reflexology from other applied therapies are; It is a healing therapy method that provides the balance strength of the body and stimulates the body's self-healing mechanism. Every part of the body has a counterpart in the hands and feet. Accordingly, reflexology to the hands and feet makes it easier to solve the problem in patients and patients. It is an easy-to-apply, no-material, medicine-assisted therapy method. Since reflexology is a method of compression and pressure, the presses on the hand reduce the stimulation of the parasympathetic and sympathetic nervous system. In the meantime, it improves blood circulation in the patient and helps one to feel peaceful and well-being. Anxiety prior to coronary angiography may lead to changes in life findings such as hypertension in patients, increased blood sugar, increased heart rate, tremor, sweating. In many studies conducted in the world and in our country related to reflexology, it was observed that the patients in the experimental group decreased their anxiety levels, breath rates, heart rates, blood pressures, milk amount of mothers and pain levels.

Inspired by these studies, the Ministry of Health of the Republic of Turkey, on the newly developing hand reflexology in our country. At the Hospital, it will be the first time to be coronary angiography for the coronary angiography, and for the first time, only femoral angiography, which is capable of filling the forms physically and mentally, without invasive procedures related to the heart. A total of 60 patients constitute the sample of the study, provided that it is planned and to accept the study. In the G-power analysis conducted to determine the sample of the study, experiment and control were calculated as 60 in total, with the sample number of both groups being 30. Since the study is a single-blind randomized clinical trial, in order to determine the randomization , a box with the names of the patients determined according to the participation criteria will be determined by the selection of the healthcare personnel responsible for the service, and the experimental and control groups. "Demographic Data Form" , "Distress Thermometer" "State Anxiety Inventory" , "Vital Signs Form" and Visual Analog Scale will be used to collect research data. The data will be taken face to face from patients who will participate in the study. The data collected from the sample group will be analyzed in program. Frequency values will be calculated to determine the distribution of categorical data, and chi-square analysis will be done and burr tables will be created. When comparing the averages of parameters containing more than two variables, variance analysis (anova) will be used and Tukey test results will be taken into consideration for significance. In repeated measurements, two-way analysis of variance (two way anova) will be used. If the research data are not normally distributed, analysis will be carried out using nonparametric tests. In this context, tests such as mann whitney u test, wilcoxon test and kruskal Wallis variance analysis will be used. In addition, the significance value of p will be considered as 0.5 for the research results to be in the 95% confidence interval .

There are not enough studies done with hand reflexology in the world and in our country. As it is an easy-to-apply, material-free therapy that can be performed under favorable conditions, it can be used to reduce anxiety before coronary angiography, to minimize stress levels and to keep changing life signs stable. Thanks to reflexology, anxiety status of the patient can be taken under control by using the internal energy of the patient without any side effects. Since reflexology is a therapy method that can be used in a wide range and shows its effect immediately, it is a method that can be used and beneficial in the field of nursing.

ELIGIBILITY:
Inclusion Criteria:

* To be applied coronary angiography for the first time waiting for coronary angiography on the same day,
* Patients over the age of 18,
* Physically and mentally patients have the ability to fill forms,
* Patients who will undergo femoral angiography, that patients agree to participate in research

Exclusion Criteria:

* Patients who do not accept the study,
* Who are physically and mentally unable to fill the forms,
* Who have sudden changes in vital signs,
* Who do not voluntarily continue

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-07-15 (Estimated); Primary Completion 2021-09-15 (Estimated); Study Completion 2022-01-15 (Estimated)

PRIMARY OUTCOMES:
Demographic form | 15 July 2021-15 October 2021three months (face to face interview)
  This form created by the researcher includes the patient's age, gender, marital status, smoking and alcohol use status, job, education level, country of origin, chronic illness, reason for angiography.

SECONDARY OUTCOMES:
Distress thermometer: | 15 July 2021-15 October 2021 three months (face to face interview) patient mark number related to distress
  It was developed by Roth et al in 1998 to determine the psychosocial distress of cancer patients.In the distress thermometer, it determines the distress level of the patient between 1 and 10 numerically.It is a simple visual scale that patients can answer even on their own.The participant expresses the distress he experiences by means of the numbers on this thermometer. 0 points indicate that the individual does not experience any distress, and 10 points indicates that the individual experiences distress at the upper limit. Distress thermometer validity and reliability study in our country in 2006. In the study, the sensitivity of the scale was 0.73 and the specificity was 0.49. In the study conducted in our country cut-off point of the scale was found to be 4.

OTHER OUTCOMES:
Vital signs | 15 July 2021-15 October 2021 three months (fever-centigrade, respiration per minute, blood pressure mmHg)
  Five vital signs, including fever, pulse, respiration, blood pressure, and pain, are measured and recorded. After the session, the vital signs of the intervention and control group are measured and recorded again.
State anxiety inventory | 15 July 2021-15 October 2021 5 minute (face to face interview) patient mark statement and give score
  It was developed by Spielberger et al. In 1970 to measure the state anxiety level of the individual.It consists of short questions and a total of 20 questions. They mark the option closest to them from the expressions such as "nothing", "a little", "a lot" and "completely" in the scale. Scores between 1 and 4 are given while answering the scale, and they can get a minimum of 20 and a maximum of 80 in total. High score indicates high anxiety, low score indicates low anxiety. At the end of the scale; 0-19 points are evaluated as no anxiety, 20-39 points as mild anxiety, 40-59 points as moderate anxiety, 60-79 points as severe anxiety, 80 points as panic.A minimum of 20 and a maximum of 80 points can be obtained from the state anxiety scale. In the scale, high scores indicate high anxiety, and low scores indicate low anxiety. In a study conducted by Oner and LeCompte (1983), the reliability of the scale was found to be between 0.94 and 0.96 for the state anxiety scale,
Visual Analog Scale | 15 July 2021-15 October 2021 three months (face to face interview) patient mark number related to pain
  The validity and reliability of the scale in our country was made in (2011); It is shown with 0 (zero) and 10 cm intervals on a ruler. On the scale, 0 (zero) means "no pain" and 10 means "worst possible pain". The patient is asked to mark the area that expresses his pain on the line. The distance marked by the patient is measured by taking the zero starting distance.

CONTACTS AND LOCATIONS:
Overall Officials: Hatice Karabuga Yakar, Study Director — Marmara University
Locations (1):
- Gebze Fatih Hospital, Kocaeli, Turkey (Türkiye)